CLINICAL TRIAL: NCT02649335
Title: To Study the Effect of Nonselective Beta Blockers in Advanced Stage Liver Disease With Ascites
Acronym: NSBB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSBB in cirrhotic ascites
Record Dates: First submitted 2015-12-05; First posted 2016-01-07 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Ascites
Keywords: Non selective beta blockers; Ascites
MeSH Terms: conditions — Ascites | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): Propranolol will be started at a dose of 40 mg and will be titrated based on pulse rate with target of 55-60 beats per minute or 20-25% reduction in heart rate and maximum tolerated dose.If any patients develop intolerable side effects, they will be withdrawn from the study.
  Interventions: Drug: Propranolol
- Endoscopic variceal ligation (EVL) (Active Comparator): Patients in EVL group will undergo regular sessions of UGIE with EVL till variceal eradication every 2- 4 weekly followed by 3 monthly for initial 6 months and 6 monthly in rest of the study period. If any patient develop acute variceal hemorrhage on follow up , will be treated inpatient with standard medical therapy (SMT) .
  Interventions: Procedure: Endoscopic variceal ligation (EVL)

INTERVENTIONS:
Drug: Propranolol — Propranolol will be started at a dose of 40 mg and will be titrated based on pulse rate with target of 55-60 beats per minute or 20-25% reduction in heart rate and maximum tolerated dose.If any patients develop intolerable side effects, they will be withdrawn from the study
  Arms: Propranolol
Procedure: Endoscopic variceal ligation (EVL) — Patients in EVL group will undergo regular sessions of UGIE with EVL till variceal eradication every 2- 4 weekly followed by 3 monthly for initial 6 months and 6 monthly in rest of the study period. If any patient develop acute variceal hemorrhage on follow up , will be treated inpatient with standard medical therapy(SMT) .
  Arms: Endoscopic variceal ligation (EVL)

SUMMARY:
Cirrhosis is the leading cause of death in India and worldwide and leading causes in developed world include alcoholic liver disease, hepatitis C, and more recently, non-alcoholic fatty liver disease (NAFLD), non-alcoholic steatohepatitis (NASH). As cirrhosis advances, portal hypertension develops, resulting in complications such as ascites, hepatic encephalopathy, and variceal hemorrhage.

Ascites is the most common major complication of cirrhosis, occurring in 50-60% of patients within ten years of diagnosis . Development of ascites is an ominous landmark in disease progression as 15% of patients with ascites will die within 1 year, and 44% within 5 years. Less than 10% patients develop refractory ascites and is associated with a poor prognosis with a high mortality, approximately 50% within 6 months and 75% at 1 year with the median survival approximately 6 months . Refractory ascites occurs as a result of splanchnic vasodilatation and maximal activation of the sympathetic nervous system (SNS) and the renin - aldosterone system (RAAS) . The therapeutic options available for these patients are serial therapeutic paracentesis, liver transplantation and trans jugular intrahepatic portosystemic shunts .The model for end stage liver disease( MELD) score predicts survival in patients with cirrhosis . However, other factors in patients with cirrhosis and ascites are also associated with poor prognosis, including low mean arterial pressure; low serum sodium, low urine sodium, and high Child-Pugh score .

Variceal bleed is the most dreaded complication of cirrhosis and screening endoscopic is recommend in these patients. About 60% of patients with decompensated cirrhosis have varices at the time of diagnosis. Majority of these patients will require non selective beta blockers (NSBB) as standard of care as primary or secondary prophylaxis in prevention of variceal hemorrhage. NSBB reduce portal pressure by decreasing cardiac output and by producing splanchnic vasoconstriction.. Endoscopic variceal band ligation (EVL) is another modality of treatment of esophageal varices and meta-analysis showed EVL to be associated with significantly lower incidence of first variceal hemorrhage without differences in mortality compared to NSBB. NSBB also has shown to improve survival in these patients with nonhemodynamic effects. Some of the patients may progress to end stage liver disease characterized by the development of refractory ascites and other complications.

Most of the studies of NSBB comparing to EVL for primary/secondary prevention of variceal hemorrhage included patients of predominantly child A/B cirrhosis with variable number with ascites without any mention of ascites grading and some of trials excluded patient's with refractory ascites. These patients with ascites received diuretics and salt restricted diet as standard of care. However none of these studies mentioned about control of ascites and survival benefit in patients with advanced stage (child B and C) cirrhosis with ascites .In recent years the role of NSBB for prevention of variceal hemorrhage in refractory ascites patients has been questioned because of the deleterious effect on survival.However the use of NSBB in end stage liver disease has shown mixed results and controversial.

Therefore this study is being planned to know the effects of NSBB in advanced stage liver disease patients with ascites and varices in preventing variceal hemorrhage ,effect on ascites and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis of any etiology with grade 2 ascites including refractory patients and varices/variceal hemorrhage requiring prophylaxis
2. Cirrhosis diagnosed by clinical, analytical, and ultrasonographic findings or available histological findings
3. Both inpatient and outpatient
4. Child B or C status

Exclusion

1. Active infection or recent infection < 2 weeks
2. Hepatic encephalopathy grade 2 or higher
3. Renal dysfunction at the time of inclusion
4. Presence of hepatocellular carcinoma or portal vein thrombosis
5. Active alcoholism
6. Pregnancy
7. HIV infection
8. Severe heart, respiratory or contraindications for beta blockers(severe chronic obstructive pulmonary disease, severe asthma, severe insulin-dependent diabetes mellitus, bradyarrhythmia)
9. Not giving consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Survival | Upto 48 weeks
  It is a categorical variable-patient dead/alive

SECONDARY OUTCOMES:
Acute kidney injury (AKI) | Upto 48 weeks
  Occurence of AKI will be noted in each group during 48 weeks follow up. The event, AKI is defined as Increase in sCr ≥0.3 mg/dl (≥26.5 μmol/L) within 48 hours; or,A percentage increase sCr ≥50% from baseline which is known, or presumed, to have occurred within the prior 7 days during study period. AKI will be treated accordingly.
Spontaneous bacterial peritonitis | 1 year
  The diagnosis is based on neutrophil count in ascitic fluid of >250/mm3 as determined by microscopy. Incidence will be noted at each follow up
Hepatorenal syndrome( HRS) | 1 year
  HRS is defined as the occurrence of renal failure in a patient with advanced liver disease in the absence of an identifiable cause of renal failure. Criteria for the diagnosis include-
  * Cirrhosis with ascites
  * Serum creatinine >1.5 mg/dl (133 lmol/L)
  * Absence of shock
  * Absence of hypovolemia as defined by no sustained improvement of renal function (creatinine decreasing to <133 lmol/L) following at least 2 days of diuretic withdrawal (if on diuretics), and volume expansion with albumin at
    1 g/kg/day up to a maximum of 100 g/day
  * No current or recent treatment with nephrotoxic drugs
  * Absence of parenchymal renal disease as defined by proteinuria <0.5 g/day, no microhaematuria (<50 red cells/high powered field), and normal renal ultrasonography.
  Incidence of HRS will be noted at each follow up.
Control of ascites | Upto 48 weeks
  Control of ascites will be assesed by clinical examination in each follow up and response to therapy will be defined as follows:
  1. Complete Response - Elimination of ascites
  2. Partial Response- Presence of ascites not requiring paracentesis.
  3. Absence of response - Persistence of ascites requiring paracentesis
  This parameter will be noted during follow up.
Incidence of variceal hemorrhage in each group | 1 year
  Occurence of variceal hemorrhage during follow up period will be noted
Incidence of Paracentesis induced circulatory dysfunction (PICD) in different groups during LVP | Upto 48 weeks
  PICD is defined as Increase in plasma renin activity of >50% of the pretreatment value on day 7 after each large volume paracentesis.

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, MD,DM, Principal Investigator — Professor of Hepatology,PGIMER,Chandigarh
Locations (1):
- Department of Hepatology,Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Derived] Singh V, Kumar P, Verma N, Vijayvergiya R, Singh A, Bhalla A. Propranolol vs. band ligation for primary prophylaxis of variceal hemorrhage in cirrhotic patients with ascites: a randomized controlled trial. Hepatol Int. 2022 Aug;16(4):944-953. doi: 10.1007/s12072-022-10361-4. Epub 2022 Jun 7. PMID 35672572